CLINICAL TRIAL: NCT06669299
Title: The Value of Late Non-Invasive Programmed Stimulation (NIPS) in the Setting of Ventricular Tachycardia (VT) Ablation to Guide the Subsequent VT Therapeutic Strategies: a Prospective Randomized Multicenter Study
Brief Title: Non-Invasive Programmed Stimulation (NIPS) to Guide the Subsequent VT Therapeutic Strategies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Dr. Paolo Della Bella, MD, IRCCS Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIPS
Record Dates: First submitted 2024-10-21; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Ventricular Tachycardia (VT)
Keywords: Ventricular Tachycardia, VT, Non-Invasive Programmed Stimulation, NIPS, ICD, Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Amiodarone; Sotalol; Mexiletine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): AAD therapy
  Interventions: Drug: Antiarrhythmic Drug Therapy (amiodarone, sotalol, or mexiletine)
- Group 2 (Experimental): Re-Do ablation procedure
  Interventions: Procedure: Re-Do ventricular tachycardia ablation

INTERVENTIONS:
Procedure: Re-Do ventricular tachycardia ablation — 1. Programmed ventricular stimulation (PVS); 2. Mapping during Sinus Rhythm (SR) or right ventricular pacing in pacing dependent patients; 3. Late Potentials identification; 4. VT(s) induction with diastolic pathway mapping when possible; 5. Catheter Ablation in SR or, at the operator's discretion, in VT if tolerated by the patient; 6. If VT is not inducible or the diastolic pathway is not mappable, a substrate ablation approach will be performed. 7. PVS is repeatedly attempting to reinduce VT after completing; 8. Endpoint: non-inducibility of any VT.
  Arms: Group 2
Drug: Antiarrhythmic Drug Therapy (amiodarone, sotalol, or mexiletine) — The patients with a positive NIPS already on antiarrhythmic drugs (AAD) before the index procedure will re-start the original antiarrhythmic therapy. Patients who were not on AAD will start a new drug at the operator's discretion (amiodarone, sotalol, or mexiletine) according to clinical practice.
  Arms: Group 1

SUMMARY:
The aim of this study is to define the importance of non-invasive programmed stimulation (NIPS) in risk stratification of ventricular tachycardia (VT) recurrence after catheter ablation and to determine the optimal treatment strategy. The primary objective is to establish whether a new VT ablation based on NIPS inducibility will reduce the risk of VT recurrence compared to antiarrhythmic drug therapy.

DETAILED DESCRIPTION:
The value of non-invasive programmed ventricular stimulation (NIPS) in the setting of ablation of ventricular tachycardia (VT) in patients with structural heart disease has been the object of studies in the last decade.

The technique is based on the feature, uniformly available in the Implantable Cardioverter-Defibrillator (ICD), to perform a complete programmed stimulation study from the apex of the right ventricle to assess the inducibility of ventricular tachycardia, similar to what is routinely performed during an invasive electrophysiology procedure. Data from our group indicate that 26% of patients who were non-inducible (apparent success) at the end of the ablation session become re-inducible to ventricular tachycardia at "late" NIPS (day 6). This finding, possibly related to partial recovery of conduction within the treated area, had prognostic significance, as it was associated with a 6-fold increased risk of VT recurrence at follow-up.

Recently Muser et al. reported similar findings (45/216 -21% of patients had clinical VT induced) with "late" NIPS performed on day 3. However, within this group of patients, the VT recurrence rate was significantly lower in those who had undergone, based on this finding, a re-do VT ablation as compared to those treated conservatively (rec in 1/11 of the Re-do ablation group, 9% vs. 24/34 in the conservative treatment group, 71%, p<0.01).

These data, however, originated from a retrospective observational analysis, where the indication of ablation was based on empirical physician preference.

No prospective randomized data compare the conservative attitude versus performing a new ablation in subjects who did not obtain a stable result after the first one. Therefore, this randomized multicenter clinical study aims to evaluate whether the repetition (Re-Do) of VT ablation process is superior to conservative medical therapy for reducing VT recurrences on post-procedural NIPS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an implanted ICD (all brands)
* Patients who underwent a successful (non-inducibility of any VT) Ventricular Tachycardia Ablation procedure, the "index procedure", supported by EnSite Precision or CARTO 3D mapping systems for the following etiologies: previous MI, myocarditis, ARVD, IDCM.
* Induction of monomorphic VT at NIPS 3-7days after a successful index procedure
* Age 18 years or more
* Able to provide an informed consent to participate to the study and available to respect the assessments described in the protocol.

Exclusion Criteria:

* Inducible VT after index procedure
* Contraindication to anticoagulants
* Presence of thrombi
* Presence of Mitral and Aortic prosthetic valve
* Recent (<3 months) myocardial infarction or unstable angina or Coronary Artery Bypass
* Pregnant or nursing
* Ventricular Tachycardia caused by reversible pathology
* < 1 Year life expectancy according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
VT recurrence free survival rate | 12 months after the procedure
  Compare the efficacy on the reduction of VT recurrence of a NIPS-based Re-Do VT ablation versus antiarrhythmic drug therapy

SECONDARY OUTCOMES:
Number of ICD shocks | Procedural, periprocedural, 6 and 12 months after procedure
Proportion of patients with VT storm | Procedural, periprocedural, 6 and 12 months after procedure
Rate of subsequent hospitalization for VT recurrence/HF. | Procedural, periprocedural, 6 and 12 months after procedure
Cardiac mortality | Procedural, periprocedural, 6 and 12 months after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Arrhythmology and Electrophysiology unit, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Della Bella P, Peretto G, Paglino G, Bisceglia C, Radinovic A, Sala S, Baratto F, Limite LR, Cireddu M, Marzi A, D'Angelo G, Vergara P, Gulletta S, Mazzone P, Frontera A. Bipolar radiofrequency ablation for ventricular tachycardias originating from the interventricular septum: Safety and efficacy in a pilot cohort study. Heart Rhythm. 2020 Dec;17(12):2111-2118. doi: 10.1016/j.hrthm.2020.06.025. Epub 2020 Jun 26. PMID 32599177
- [Background] Irie T, Yu R, Bradfield JS, Vaseghi M, Buch EF, Ajijola O, Macias C, Fujimura O, Mandapati R, Boyle NG, Shivkumar K, Tung R. Relationship between sinus rhythm late activation zones and critical sites for scar-related ventricular tachycardia: systematic analysis of isochronal late activation mapping. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):390-9. doi: 10.1161/CIRCEP.114.002637. Epub 2015 Mar 4. PMID 25740836
- [Background] Muser D, Hayashi T, Castro SA, Supple GE, Schaller RD, Santangeli P, Arkles J, Kumareswaran R, Nazarian S, Deo R, Lin D, Dixit S, Epstein AE, Callans DJ, Marchlinski FE, Frankel DS. Noninvasive Programmed Ventricular Stimulation-Guided Management Following Ventricular Tachycardia Ablation. JACC Clin Electrophysiol. 2019 Jun;5(6):719-727. doi: 10.1016/j.jacep.2019.03.007. Epub 2019 May 1. PMID 31221360
- [Background] Oloriz T, Baratto F, Trevisi N, Barbaro M, Bisceglia C, D'Angelo G, Yamase M, Paglino G, Radinovic A, Della Bella P. Defining the Outcome of Ventricular Tachycardia Ablation: Timing and Value of Programmed Ventricular Stimulation. Circ Arrhythm Electrophysiol. 2018 Mar;11(3):e005602. doi: 10.1161/CIRCEP.117.005602. PMID 29545359